CLINICAL TRIAL: NCT06364553
Title: Esophageal Self-expandable Metal Stent for Malignant Strictures: a Safety and Efficacy Study
Acronym: ENTRANCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Peter Siersema, Prof. dr., Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL86416.078.24
Record Dates: First submitted 2024-04-03; First posted 2024-04-15 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Oesophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Esophageal self-expandable metal stent (Other): Esophageal self-expandable metal stent
  Interventions: Device: Esophageal self-expandable metal stent

INTERVENTIONS:
Device: Esophageal self-expandable metal stent — The Leufen Esophageal aixstent ® (Leufen Medical GmbH) is indicated for the treatment of malignant esophageal strictures and postoperative stenosis. It is comprised of two components: an implantable metallic stent and the delivery system. After the procedure, the stent remains at the intended location, within the patient while the delivery system is removed.

SUMMARY:
A single center prospective observational non-randomized clinical study to assess the safety and efficacy of placement of a new esophageal self-expandable metal stent (SEMS) for palliation of patients with malignant dysphagia.

DETAILED DESCRIPTION:
Objective: To assess the safety and efficacy of placement of a new esophageal self-expandable metal stent (SEMS) for palliation of patients with malignant dysphagia.

Study design: Single center prospective observational non-randomized clinical study.

Study population: A total of 20 patients with malignant dysphagia will be included. Sample size calculation does not apply for this type of study. Outcome of the study (efficacy and safety) will be compared to our historic esophageal stent database, including over 1000 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with dysphagia due to a non-curable malignant obstruction of the esophagus or esophagogastric junction including extrinsic malignant compression and recurrence in post-esophagectomy patients;
* Requiring treatment for dysphagia (Ogilvie score of 2-41);
* Life expectancy of less than 12 months;
* Written informed consent;
* Age ≥ 18 years.

Exclusion Criteria:

* Stenosis after laryngectomy;
* Distance between the upper edge of the stent less than 2 cm from the upper esophageal sphincter;
* Tumor length of more than 14 cm;
* Previous stent placement for the same condition;
* Coagulopathy (not corrected prior to stent placement);
* Patients with eosinophilic esophagitis or an esophageal motility disorder;
* Nickel titanium (Nitinol) allergy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Complication: incidence of perforation | 6 months
  The complication perforation during stent placement and during follow-up will be measured using patient anamneses and if necessary upper endoscopy and described as present yes or no. After all patients are included, the incidence can be described as percentage.
Complication: incidence of hemorrhage | 6 months
  The complication hemorrhage will be measured during stent placement and follow-up using patient anamneses and if necessary with an upper endoscopy and described as present yes or no. After all patients are included, the incidence can be described as percentage.
Complication: incidence of fistula formation | 6 months
  The complication fistula formation will be measured during stent placement and during follow-up using patient anamneses and if necessary with an upper endoscopy and is described as present yes or no. After all patients are included, the incidence can be described as percentage.
Complication: incidence of gastroesophageal reflux | 6 months
  The complication gastroesophagel reflux will be measured after stent placement with the use of patient anamneses and will be described as present yes or no. After all patients are included, the incidence can be described as percentage.
Complication: incidence of stent migration | 6 months
  The complication stent migration will be measured using a new upper endoscopy in case there is recurrent dysphagia (measured with the Ogilvie Dysphagia score from 0 = no dysphagia to 4 = inability to swallow food or liquids, so the higher te score, the worse the outcome) and described as present yes or no. After all patients are included, the incidence can be described as percentage.
Efficacy: clinical outcome | 6 months
  The clinical outcome will be measured using the Ogilvie Dysphagia Score to determine whether recurrent dysphagia is present after stent placement during follow-up or until death. The Ogilvie Dysphagia Score is a score ranging from 0 = no dysphagia to 4 = inability to swallow any food or liquids, so the higher te score, the worse the outcome.
Efficacy: incidence of patients receiving technical successful stent placement | 1 day, during stent placement
  Technical successful stent placement will be measured during stent placement whether the stent is in the correct position (covering the whole stenosis) and is described as yes or no. After all patients are included, the incidence can be described as percentage.

SECONDARY OUTCOMES:
Incidence of recurrent dysphagia | 6 months
  Recurrent dysphagia will be asked from the patient and will be measured with the Ogilvie Dysphagia score (ranging from 0 = no dysphagia to 4 = inability to swallow any food or liquids, so the higher te score, the worse the outcome). After all patients are included, the incidence can be described as percentage.
Pain related to esophageal stent (placement) | 6 months
  Pain related to esophageal stent (placement) measured daily using a patient diary which scores the Visual Analogue Scale (ranging from 0 = no pain to 10 = the worst pain imaginable, so the higher the score, the worse the outcome) during the first two weeks, after this every 4 weeks a telephone call with the patient will be held to discuss pain using the Visual Analogue Scale as well until death/stent removal, or until a maximum of 6 months follow-up)
Overall survival | 6 months
  Overall survival measured in days

OTHER OUTCOMES:
Patient characteristic: age | 1 day, at stent placement
  Patient age at baseline, so at the day of stent placement, measured in years
Patient characteristic: gender | 1 day, at stent placement
  Patient gender at baseline, at the day of stent placement, measured as male or female
Patient characteristic: tumor location | 1 day, during stent placement
  Location of the tumor in the esophagus, measured in cm from incisors during stent placement
Patient characteristic: tumor histology | 1 day, checking PA records
  Histology of the tumor in the esophagus, measured from biopsy results from upper endoscopies perfomed prior to the stent placement
Stent characteristic: length of the stent | 1 day, during stent placement
  Length of the stent, determined during stent placement in millimeters
Stent characteristic: diameter of the stent | 1 day, during stent placement
  Diameter of the stent, determined during stent placement in millimeters
Patient characteristic: prior radiotherapy | 1 day, before stent placement
  Determining whether patient received radiotherapy prior to the stent placement, described as yes or no
Patient characteristic: prior chemotherapy | 1 day, before stent placement
  Determining whether patient received chemotherapy prior to the stent placement, described as yes or no

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands